CLINICAL TRIAL: NCT04590261
Title: Myeloid Cells in Patients With Covid-19 Pneumonia
Acronym: MyeloidCovid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APHP201138; 2020-A02700-39 (Other: IDRCB)
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Covid-19; SARS-Cov2
Keywords: Covid-19; Neutrophils; Dendritic cells; Monocytes; Macrophages; Interferons; Nasal mucosa; Peripheral blood; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Other): Former mild SARS-Cov2 Pneumonia, 2 to 12 moths before, ≤ 5 L/mn Oxygen treatment
  Interventions: Other: Blood sampling; Other: Nasal Brushing
- Group 2 (Other): Former severe SARS-Cov2 Pneumonia, 2 to 12 moths before, > 5 L/mn Oxygen treatment
  Interventions: Other: Blood sampling; Other: Nasal Brushing
- Group 3 (Other): Physician examination in the Pneumology ward, Cochin Hospital
  Interventions: Other: Blood sampling; Other: Nasal Brushing
- Group 4 (Other): Current hospitalization for Sars-Cov2 Pneumonia at Cochin Hospital
  Interventions: Other: Blood sampling; Other: Nasal Brushing

INTERVENTIONS:
Other: Blood sampling — Peripheral Blood sampling, 25 mL
Other: Nasal Brushing — Nasal Brushing, facultative

SUMMARY:
The purpose of this study is to analyze in depth the relationship of myeloid cell subpopulations during infection by Severe acute respiratory syndrome coronavirus 2 (SARS-Cov2), the virus mediating Covid-19. Myeloid cells include neutrophils, monocytes and dendritic cells, each divided into subpopulations with different functions in immune defense and immune pathologies.

The study is based on the following hypotheses:

* Infection and the interferon response to infection may induce hyperactive or immunosuppressive differentiation of myeloid cells, that may be treated by specific inhibitors.
* Some myeloid cell subpopulations currently identified in our laboratories might be markers for Covid-19 prognosis.
* Alternative receptors may be present on myeloid cells, inducing the cytokine storm, a target for therapy.
* The expression of Interferon (IFN) receptor and IFN responding genes on myeloid cells and on respiratory epithelial cells may correlate with prognosis and indicate potential treatment targets.
* Interferon responses are known to be skewed during Covid-19, but some IFN subtype polymorphisms may correlate with prognosis and these subtypes migt be supplemented or inhibited for therapy.

DETAILED DESCRIPTION:
Infection by SARS-Cov2 drives to pneumonia in most cases, 30 percent of which require hospitalization in a pneumology ward, among which 30 percent with severe acute respiratory syndrome (SARS) must go to critical care units, with a high mortality rate.

This infection drives a strong cytokine response. In patients developing SARS, a profound, paradoxical defect in IFN alpha and in the expression of genes responding to IFN alpha was discovered. IFNs are strong anti-viral proteins, used for the treatment of viral hepatitis. Type I IFNs, including IFN alpha, have ubiquitous receptors on almost every cell type. Type III IFNs, or IFN lambda, have a more restricted receptor expression, including on neutrophils. Their polymorphisms were already related to the prognosis of another ribonucleic acid (RNA) virus with mucosal entry, hepatitis C virus (HCV), especially in people with African origins.

Coronaviruses responsible for the previous SARS-Cov or Middle East respiratory syndrome coronavirus (MERS-Cov) epidemics induce a defective IFN signal transduction. Many other viral infection lead to desensitization. Moreover, IFN alpha by itself can lead to defective antiviral responses. At the immune cell level, lymphopenia with an increased neutrophil/lymphocyte ratio were noted in severe SARS-Cov2 case. New subpopulations of neutrophils have been characterized by phenotypic and proteomic studies, with inflammatory or suppressive functions.

It will be important to know if

* hyperactive or immunosuppressive myeloid cell differentiation is caused by SARS-Cov2 and can be inhibited specifically.
* some myeloid subpopulations
* correlate with the prognosis of the disease,
* myeloid cells have alternative receptors for SARS-Cov2,
* some IFN polymorphisms may correlate with prognosis and might be supplemented or inhibited for therapy.

The answers will be obtained through the primary and secondary outcome measures, as described below.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Sex : male or female
* French Social Security insurance
* Information and consent dated and signed *
* Group 1 : inclusion 2 to 12 months after hospitalization for Covid-19 pneumonia with mild severity (oxygen treatment ≤5L/mn);
* Group 2 : 2 to 12 months after hospitalization for Covid-19 pneumonia with high severity (oxygen treatment >5L/mn);
* Group 3 : external visit at Cochin Hospital, age- and sex -matched with Groups 1, 2, 4.
* Group 4 : inclusion during hospitalization for Covid-19, within the first month of symptoms.

Exclusion Criteria:

* Tuberculosis or other evolutive bacterial infection
* Chronic evolutive viral Infections (Hepatitis B or C, HIV)
* Ongoing chemotherapy or radiotherapy
* Participation in another research protocol with current exclusion period at the time of pre-inclusion (possible inclusion in an observational study
* Vulnerable person (pregnant, parturient woman, breastfeeding woman, person Under tutorship, person under arrest through judiciary or administrative decision )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Myeloid cell sub-population phenotype | Month zero-month 36
  Cytometric analysis of surface and intracellular molecules to identify myeloid cell sub-populations and define their function in vivo

SECONDARY OUTCOMES:
Myeloid cell functions | Month zero-month 36
  Cell culture and cytometric and analyte analysis of their functions, including IFN production
Myeloid cell transcriptomic and proteomic study | Month zero-month 36
  Transcriptomic and proteomic analysis of the functions of myeloid cell subtypes
Transcriptomic study of nasal epithelial cells | Month zero-month 36
  Single cell RNA sequencing of the nasal brush products
Plasma analyte concentration measurement | Month zero-month 36
  High sensitivity detection by state-of-the art ELISA type methods

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Régis Burgel, MD, PhD, Principal Investigator — Cochin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Team Niedergang — https://www.institutcochin.fr/la-recherche/3i/equipe-niedergang